CLINICAL TRIAL: NCT02726451
Title: A Post-Market, Randomized, Placebo-Controlled Study to Assess the Efficacy of Cosmeceutical Therapy in Subjects Undergoing Full Facial Rejuvenation
Brief Title: A Study to Examine the Effects of Cosmeceutical Therapy in Subjects Undergoing Full Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PCA-SD-01
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Facial Rejuvenation With Neurotoxins and/or Hyaluronic Acid Fillers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basic Skin Care (Placebo Comparator): Subjects use a basic skin care regimen.
  Interventions: Other: Basic Skin Care
- Active Skin Care (Active Comparator): Subjects use the Sensi Peel®, Rejuvenating Serum, and C&E Strength Max skin care products in additional to a basic skin care regiment.
  Interventions: Other: Active Skin Care

INTERVENTIONS:
Other: Basic Skin Care — Facial Wash, Hydrator Plus Broad Spectrum SPF 30, and Rebalance skin care products (PCA SKIN®)
  Other Names: Group A
  Arms: Basic Skin Care
Other: Active Skin Care — Sensi Peel®, Rejuvenating Serum, and C&E Strength Max skin care products (PCA SKIN®) in addition to the Facial Wash, Hydrator Plus Broad Spectrum SPF 30, and Rebalance skin care products (PCA SKIN®)
  Other Names: Group B
  Arms: Active Skin Care

SUMMARY:
The primary objective of this study is to determine the efficacy of Sensi Peel®, Rejuvenating Serum, and the C&E Strength Max skin care products in subjects who undergo full facial rejuvenation, with a botulinum neurotoxin A and/or hyaluronic acid filler, in improving the appearance of the skin, patient satisfaction with aesthetic appearance, and the projected first impressions.

The secondary objective of this study is to examine patient satisfaction with the continuous use of Sensi Peel®, Rejuvenating Serum, and the C&E Strength Max products.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female between the ages of 21 and 60;
* Subject requires a full facial rejuvenation with a HA soft tissue filler and/or botulinum neurotoxin, per judgment of the PI or designee;
* Subject is willing and able to provide written informed consent prior to the performance of any study related procedure;
* Subject is willing and able to comply with the protocol requirements; and
* Subject is willing and able to provide written photo consent and adhere to the photography and video procedures such as removal of jewelry and makeup.

Exclusion Criteria:

* Subjects who have received any facial filler in the 12-month or neurotoxin treatments in the 4-month period prior to enrollment;
* Previous treatment with any resurfacing facial aesthetic procedure (e.g. deep chemical peeling and laser treatments) within the 12-month period prior to enrollment;
* Previous treatment with photo rejuvenation therapy within the 6-month period prior to enrollment;
* Subjects who plan to undergo facial cosmetic surgery or any aesthetic procedure (e.g. neurotoxins, dermal fillers, laser treatments, and chemical peels), which are not specified in this protocol, during the course of the study;
* A known allergy or sensitivity to any component of the study ingredients;
* Use of systemic steroids or anticoagulation medications;
* Subjects with a history of bleeding disorders;
* Subjects with severe allergies manifested by a history of anaphylaxis or presence of multiple severe allergies;
* Subjects with hypersensitivity to botulinum neurotoxin;
* Subject with allergies to gram positive bacterial proteins;
* Sensitivity to sulfides;
* Subjects with allergy to cow's milk protein;
* Subjects with previous history of sensitivity to amide type local anesthetics;
* Subject with surgical alterations to the facial anatomy or marked facial asymmetry;
* Inflammation or infection at the injection site(s);
* Subjects with a history of eyelid or eyebrow ptosis;
* Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin;
* Subjects with neuromuscular disorders;
* Use of anticholinergic, aminoglycosides or other agents that interfere with neuromuscular transmission (e.g., curare-like agents), or muscle relaxants;
* Subjects with immunodeficiencies such as HIV, lupus, scleroderma, and systemic infections;
* Pregnant, nursing, or sexually active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence);
* Current history of chronic drug or alcohol abuse;
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study product;
* Subjects who, in the investigator's opinion, have a history of poor cooperation, non-compliance with medical treatment, or unreliability; and
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11-07 (Actual); Study Completion 2016-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Basic Skin Care | Active Skin Care
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic Skin Care | Active Skin Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 54.3 [41 to 68] | 54.3 [41 to 68] | 54.3 [41 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: C-GAIS by the PI or Designee
Description: Global aesthetic improvement in subjects is assessed by the PI/designee using the Global Aesthetic Improvement Scale (C-GAIS).
  Clinical-Global Aesthetic Improvement Scale (C-GAIS):
  3 (Very Much Improved) 2 (Much Improved)
  1 (Improved) 0 (No change)
  -1 (Worse)
  Scores closer to 3 show a more favorable outcome Scores closer to -1 show a less favorable outcome
Time Frame: Approximately 3 months from the baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basic Skin Care | Active Skin Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Visit 7 | 1.22 (0.441) | 2.13 (0.835)
  Visit 8/9 | 1.75 (0.886) | 2.75 (0.787)

2. Primary Outcome: SQA by the PI or Designee
Description: The quality of subjects' skin is assessed by PI/designee using the Skin Quality Assessment (SQA)
  Skin Quality Assessment (SQA):
  Tone (dyschromia) 0 - severe unevenness
  1- moderate to severe unevenness 2 - moderate unevenness 3 - mild unevenness 4 - even
  Elasticity (Firmness) 0 - Very poor elasticity
  1. - poor elasticity
  2. - fair elasticity
  3. - good elasticity
  4. - firm
  Texture (Smoothness) 0 - severe
  1. - moderate to severe
  2. - moderate
  3. - mild
  4. - none
  Radiance 0 - severe dullness
  1. - moderate to severe dullness
  2. - moderate dullness
  3. - mild dullness
  4. - radiant
  All scores with a higher number indicate favorable results All scores with a lower number indicate less favorable results
Time Frame: Approximately 3 months from the baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basic Skin Care | Active Skin Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Tone - Visit 1 | 1.44 (0.527) | 1.20 (0.422)
  Tone - Visit 7 | 1.78 (0.667) | 2.75 (0.707)
  Tone - Visit 8/9 | 2.88 (0.641) | 3.14 (0.690)
  Elasticity - Visit 1 | 1.33 (0.5) | 1.30 (0.483)
  Elasticity - Visit 7 | 2.33 (0.5) | 3.25 (0.886)
  Elasticity - Visit 8/9 | 2.75 (0.707) | 3.57 (0.535)
  Texture - Visit 1 | 1.11 (0.601) | 1.10 (0.316)
  Texture - Visit 7 | 2.33 (0.5) | 3.25 (0.886)
  Texture - Visit 8/9 | 2.88 (0.835) | 3.71 (0.488)
  Radiance - Visit 1 | 0.88 (0.354) | 1.0 (.0)
  Radiance - Visit 7 | 2.25 (0.707) | 3.25 (0.886)
  Radiance - Visit 8/9 | 3.00 (0.926) | 3.71 (0.488)

3. Secondary Outcome: Face-Q by Subjects
Description: Subjects self-evaluation of their quality of skin, age-appraisal, and social and psychological assessments are performed using the Face-Q questionnaire.
  FACE-Q (Satisfaction with Skin): scored between 1-4 for 12 questions. Total score closer to 48 indicates a more favorable outcome FACE-Q (Satisfaction with Facial Appearance Overall): scored between 1-4 for 10 questions. Total score closer to 40 indicates a more favorable outcome FACE-Q (Aging Appearance Appraisal): scored between 1-4 for 7 questions. Total score closer to 28 indicates a more favorable outcome FACE-Q (Age Appraisal-VAS): scored between -15 to +15. Total score closer to -15 indicates a more favorable outcome FACE-Q (Psychological Well-Being): scored between 1-4 for 10 questions. Total score closer to 40 indicates a more favorable outcome FACE-Q (Social Function):scored between 1-4 for 8 questions. Total score closer to 32 indicates a more favorable outcome
Time Frame: Final assessment is approximately 3 months from the baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basic Skin Care | Active Skin Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Satisfaction with Skin - V5 | 3.21 (0.88) | 3.54 (0.778)
  Satisfaction with Skin - V7 | 3.27 (0.667) | 3.29 (0.787)
  Satisfaction with Skin - V8/9 | 3.6 (0.641) | 3.18 (0.690)
  Satisfaction with Facial Appearance Overall - V5 | 3.14 (0.5) | 3.13 (0.483)
  Satisfaction with Facial Appearance Overall - V7 | 3.08 (0.5) | 3.06 (0.886)
  Satisfaction with Facial Appearance Overall - V8/9 | 3.46 (0.707) | 3.1 (0.535)
  Aging Appearance Appraisal - V5 | 2.22 (0.601) | 1.79 (0.316)
  Aging Appearance Appraisal - V7 | 2.08 (0.5) | 1.88 (0.886)
  Aging Appearance Appraisal - V8/9 | 1.45 (0.835) | 1.61 (0.488)
  Age Appraisal-VAS - V5 | -2 (0.354) | -3 (0.5)
  Age Appraisal-VAS - V7 | -2.22 (0.707) | -3.13 (0.886)
  Age Appraisal-VAS - V8/9 | -5.38 (0.926) | -3.57 (0.488)
  Psychological Well-Being - V5 | 3.5 (0.568) | 3.54 (0.526)
  Psychological Well-Being - V7 | 3.52 (0.552) | 3.66 (0.59)
  Psychological Well-Being - V8/9 | 3.81 (0.699) | 3.8 (0.658)
  Social Function - V5 | 3.51 (0.553) | 3.53 (0.633)
  Social Function - V7 | 3.56 (0.878) | 3.58 (0.925)
  Social Function - V8/9 | 3.67 (0.787) | 3.57 (0.477)

4. Secondary Outcome: SSES by Subjects
Description: Changes in self-esteem is assessed using the State Self-Esteem Scale (SSES): performance, social, and appearance
  State Self-Esteem Scale (SSES): scored between 1-5 for 20 questions. Scores closer to 100 indicate a more favorable outcome
Time Frame: Final assessment is approximately 3 months from the baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basic Skin Care | Active Skin Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 80.5 (0.527) | 78.5 (0.422)
  Visit 7 | 79 (0.886) | 80 (0.707)
  Visit 8/9 | 84 (0.641) | 85 (0.690)

5. Secondary Outcome: FIQ by Blinded Evaluators
Description: The projected first impressions are assessed by blinded evaluators using the First Impression Questionnaire (FIQ).
  First Impression Questionnaire (FIQ): scored between 1-10 for 8 questions. Scores closer to 10 for each question indicate a more favorable outcome
Time Frame: At the conclusion of study assessments (approximately 3 months from the baseline visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basic Skin Care | Active Skin Care
Number analyzed (Participants) | 10 | 10
units on a scale
  Social skills - Before | 4.9525 (0.79094) | 5.0600 (0.83857)
  Social skills - After | 5.9136 (0.64010) | 6.3333 (1.67975)
  Academic Performance - Before | 5.3400 (0.83351) | 5.3900 (0.78095)
  Academic Performance - After | 6.1550 (0.48823) | 6.2800 (1.63815)
  Dating success - Before | 4.6700 (1.21824) | 5.0367 (0.99995)
  Dating success - After | 5.5470 (0.85017) | 6.1433 (1.85263)
  Occupational success - Before | 5.3350 (0.93159) | 5.5233 (0.77835)
  Occupational success - After | 6.0723 (0.57428) | 6.3967 (1.58576)
  Attractiveness - Before | 4.7225 (1.27725) | 4.9467 (1.07574)
  Attractiveness - After | 5.7758 (1.03805) | 6.0867 (1.95090)
  Financial Success - Before | 5.3025 (0.92139) | 5.3567 (0.81363)
  Financial Success - After | 6.0309 (0.61463) | 6.2467 (1.58249)
  Relationship success - Before | 5.0850 (0.96094) | 5.2167 (0.76078)
  Relationship success - After | 5.9597 (0.69371) | 6.3233 (1.70127)
  Athletic success - Before | 4.6475 (1.31627) | 4.6767 (1.03115)
  Athletic success - After | 5.4897 (0.96880) | 5.7467 (1.67741)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Basic Skin Care | Active Skin Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes